CLINICAL TRIAL: NCT01179802
Title: Magnetic Resonance Technique in the Assessment of Exercise-induced Long- and Short-Term Changes in Cardiac Function and Morphology
Brief Title: Exercise-induced Changes in Cardiac Function & Morphology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Federal Office of Sports, Switzerland (Other Government)
Responsible Party: Dr.phil.nat. Dr.sci.med. Michael Ith, Dept. of Diagnostic, Interventional and Pediatric Radiology (DIPR) University & Inselspital Bern
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KEK 005/10
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Myocardial Ischemia; Exercise; Myocardial Contraction; Myocardial Stunning; Heart Failure
MeSH Terms: conditions — Myocardial Ischemia; Motor Activity; Myocardial Stunning; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): single event of a prolonged strenuous endurance exercise (mountain marathon)
  Interventions: Other: Strenuous Endurance exercise

INTERVENTIONS:
Other: Strenuous Endurance exercise — "Jungfraumarathon": Mountain-Marathon with a length of 42km and a altitude-difference of approximately 1830meters.

SUMMARY:
Until now it has been assumed that regular endurance training has a positive influence on cardiac function and that the positive effect increases with increasing intensity. However, little is known about the effects of intense endurance stress on the heart. According to current knowledge repeated exposure to strenuous endurance activity may lead to minor but possibly irreversible damage to the heart with resultant scarring of the heart's muscle.

Within this study we attempt to find out by different analytical methods - in particular magnetic resonance imaging (MRI) and ultrasound of the heart - to what extent the heart muscle is affected by an intense endurance exercise, i.e. the "Jungfrau-Marathon", and which changes can possibly be found. Due to repeated measurements we will obtain further information on the short-term course of possible changes.

Hypotheses: A single bout of prolonged strenuous exercise (PSE) leads to transient alteration in cardiac function accompanied by the appearance of biomarkers for myocardial damage.

DETAILED DESCRIPTION:
Background

Despite the well documented cardio-protective effects of aerobic exercise of moderate intensity, short- and long-term consequences of strenuous exercise are less clear. There is increasing evidence that maintaining a high cardiac workload over a prolonged duration may result in transient impairment of cardiac function. Recent studies have also reported a transient increase in cardiac biomarkers after prolonged strenuous exercise. While in patients with cardiac disease the presence of cardiac dysfunction and increased cardiac biomarkers generally reflects myocardial damage, the impact of these observations in athletes is ill defined. It is a matter of concern whether in athletes such findings simply reflect a reversible response or whether repetitive events may lead to an accumulative cardiac damage. Traditional echocardiographic methods used to determine potential cardiac changes in morphology or function are investigator-dependent and may be subject to interference by cardiac pre- and afterload. Cardiac magnetic resonance imaging provides an investigator-independent and objective method to quantify cardiac dimensions and function. Delayed contrast enhancement MR imaging is a highly reproducible cardiovascular magnetic resonance imaging technique to directly visualize myocardial edema, necrosis and fibrosis.

Objective

To use cardiac and delayed contrast enhancement magnetic resonance imaging in combination with echocardiographic methods to quantify cardiac dysfunction after a single competitive PSE event and to study post-exercise changes in morphology and function as well as the post-exercise dynamics of specific markers of myocardial damage.

Methods

Cardiac and delayed contrast enhancement magnetic resonance imaging will be used in combination with echocardiographic methods to repetitively investigate post-exercise cardiac function and morphology in 10 elite athletes finishing the "Jungfrau Marathon". Biomarkers of myocardial damage are assessed simultaneously.

Post-exercise dynamics of the outcome parameters are followed over a minimum of 7 days after the exercise.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the Jungfraumarathon 2010
* Elite runners defined by their results in the Jungfraumarathon 2009 (not more than 4:30 h, corresponding to a delay of 90 minutes compared to the winner)

Exclusion Criteria

* Contraindication for MRI
* • History of relevant cardiac disease (including cardiomyopathies)
* coronary heart disease
* coronary abnormalities
* cardiovascular risk factors
* History of any chronic disease
* drug abuse

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Quantification of edema and/or ischemic areas with MRI | baseline
Quantification of edema and/or ischemic areas with MRI | 24h post-marathon
Quantification of edema and/or ischemic areas with MRI | 5 days post-marathon
Quantification of edema and/or ischemic areas with MRI | 8 days post-marathon

SECONDARY OUTCOMES:
anthropometric data, VO2max, resting-ECG, stress-ECG, blood analyses | at baseline
Cardiac contractility by echocardiography | 1h post-marathon
Cardiac contractility by echocardiography | 5 days post-marathon
Cardiac contractility by echocardiography | 8 days post-marathon
Cardiac contractility by echocardiography | baseline
various parameters of cardiac function and morphology assessed with MRI and echocardiography | baseline
various parameters of cardiac function and morphology assessed with MRI and echocardiography | 1h post-marathon
various parameters of cardiac function and morphology assessed with MRI and echocardiography | 1 day post-marathon
various parameters of cardiac function and morphology assessed with MRI and echocardiography | 5 days post-marathon
various parameters of cardiac function and morphology assessed with MRI and echocardiography | 8 days post-marathon
Post-exercise levels and dynamics of blood parameters indicating cardiac damage, cardiac overload , inflammation and hormonal stress response | baseline
Post-exercise levels and dynamics of blood parameters indicating cardiac damage, cardiac overload , inflammation and hormonal stress response | 1h post-marathon
Post-exercise levels and dynamics of blood parameters indicating cardiac damage, cardiac overload , inflammation and hormonal stress response | 1 day post-marathon
Post-exercise levels and dynamics of blood parameters indicating cardiac damage, cardiac overload , inflammation and hormonal stress response | 5 days post-marathon
Post-exercise levels and dynamics of blood parameters indicating cardiac damage, cardiac overload , inflammation and hormonal stress response | 8 days post-marathon

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ith, PhD, PhD/MD, Principal Investigator — Dept. of Diagnostic, Interventional and Pediatric Radiology, University Hospital Bern; Christoph Stettler, MD, Principal Investigator — Division of Endocrinology, Diabetes and Clinical Nutrition, University Hospital Bern
Locations (1):
- Dept. of Diagnostic, Interventional and Pediatric Radiology, University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Derived] Wilhelm M, Zueger T, De Marchi S, Rimoldi SF, Brugger N, Steiner R, Stettler C, Nuoffer JM, Seiler C, Ith M. Inflammation and atrial remodeling after a mountain marathon. Scand J Med Sci Sports. 2014 Jun;24(3):519-25. doi: 10.1111/sms.12030. Epub 2012 Dec 18. PMID 23253265